CLINICAL TRIAL: NCT00277771
Title: Improving Self-Monitoring in Weight Loss With Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lora Burke (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Lora Burke, Professor of Nursing and Epidemiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0507098; 1R01DK071817-01 (NIH)
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Obesity; Overweight
Keywords: technology in weight loss; standard behavioral therapy for obesity
MeSH Terms: conditions — Obesity; Overweight | interventions — Serum Bactericidal Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Standard behavioral treatment (SBT) for weight loss — Participants attend group sessions where they learn about healthy eating and exercise. They are asked to self-monitor all calories consumed (food and drink) and all calories expended through exercise. Standard paper diaries are used for self-monitoring.
Behavioral: SBT for weight loss using a PDA — Participants attend group sessions where they learn about healthy eating and exercise. They are asked to self-monitor all calories consumed (food and drink) and all calories expended through exercise. Personal Digital Assistants (PDAs) are used for self-monitoring.
Behavioral: SBT for weight loss using a PDA with feedback messages — Participants attend group sessions where they learn about healthy eating and exercise. They are asked to self-monitor all calories consumed (food and drink) and all calories expended through exercise. Personal Digital Assistants with a customized feedback program are used for self-monitoring.

SUMMARY:
We propose to conduct a randomized study of standard behavioral weight-loss treatment to test if using an electronic diary with or without tailored feedback will improve adherence to self-monitoring and subsequently improve weight loss. Subjects will be randomly assigned to different methods to self-monitor food and exercise habits: (1) use of the traditional paper diary , (2) use of a personal digital assistant (PDA), or (3) use of a personal digital assistant that also provides daily feedback.

DETAILED DESCRIPTION:
The prevalence of obesity, a major chronic health problem that is an independent risk factor for coronary heart disease (CHD), continues to increase at an alarming rate. Although weight control research has significantly improved short-term treatment success, long-term weight loss maintenance has lagged behind. Research has demonstrated a consistent relationship between self-monitoring eating and physical activity habits and success in weight loss as well as in maintenance of weight loss. However, the methods primarily used for self-monitoring continue to be the paper diary (PD), which is time consuming and burdensome. Moreover, PDs do not permit immediate external feedback to support and motivate the individual. Emerging technologies could improve self-monitoring and weight loss treatment. However, the use of these technological advances, such as a personal digital assistant (PDA), has not been studied in weight loss treatment. The primary aim of this behavioral weight loss treatment study is to determine if self-monitoring of daily eating and physical activity habits using a PDA, with or without a tailored feedback intervention, is superior to using a PD in terms of promoting and maintaining short- and long-term weight loss. Secondary aims include comparing the effect of treatment group assignment on adherence to self-monitoring and on risk factors for CHD (lipids, glucose, insulin, C-reactive protein). We propose to enroll 198 subjects and randomize them to one of three treatment groups that will use different methods to self-monitor eating and physical activity habits: (1) use of the traditional PD with delayed written feedback, (2) use of a PDA with limited feedback on daily targets, or (3) use of a PDA with limited feedback on daily targets plus receive daily, subject-tailored feedback messages via the PDA. The proposed study includes prolonged (24 months) supervision of self-management with three important components: self-monitoring, feedback, and ongoing contact. Subjects will complete assessments at baseline, 6, 12, 18, and 24 months. This innovative study will provide information on the efficacy of combining technological advances with proven behavioral strategies.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 59 years
2. BMI ≥ 27 and ≤ 43
3. willing to be randomized to one of the three treatment conditions
4. successful completion of screening

   * Note that although residing in Western Pennsylvania is not an explicit eligibility criterion, participants are asked to travel to the University of Pittsburgh frequently.

Exclusion Criteria:

1. presence of an eating disorder
2. current serious illness or unstable condition requiring physician-supervised diet and exercise including a glucose level above 125 at baseline
3. physical limitations precluding ability to exercise
4. pregnant or planning to become pregnant in the next 24 mos
5. under current treatment for a psychological disorder
6. reported alcohol intake of 4 drinks/day or more
7. current or recent (past 6 mos) participation in a weight-loss program or use of weight-loss medication
8. planning an extended vacation, absence, or relocation within the next 24 mos

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2006-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Weight Change | Measured every 6 months

SECONDARY OUTCOMES:
Adherence to self-monitoring | Measured throughout the study
Coronary heart disease risk factors (lipid, glucose, insulin) | Measures annually

CONTACTS AND LOCATIONS:
Overall Officials: Lora E. Burke, PhD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Goode RW, Ye L, Sereika SM, Zheng Y, Mattos M, Acharya SD, Ewing LJ, Danford C, Hu L, Imes CC, Chasens E, Osier N, Mancino J, Burke LE. Socio-demographic, anthropometric, and psychosocial predictors of attrition across behavioral weight-loss trials. Eat Behav. 2016 Jan;20:27-33. doi: 10.1016/j.eatbeh.2015.11.009. Epub 2015 Nov 14. PMID 26609668
- [Derived] Turk MW, Elci OU, Wang J, Sereika SM, Ewing LJ, Acharya SD, Glanz K, Burke LE. Self-monitoring as a mediator of weight loss in the SMART randomized clinical trial. Int J Behav Med. 2013 Dec;20(4):556-61. doi: 10.1007/s12529-012-9259-9. PMID 22936524
- [Derived] Burke LE, Styn MA, Sereika SM, Conroy MB, Ye L, Glanz K, Sevick MA, Ewing LJ. Using mHealth technology to enhance self-monitoring for weight loss: a randomized trial. Am J Prev Med. 2012 Jul;43(1):20-6. doi: 10.1016/j.amepre.2012.03.016. PMID 22704741